CLINICAL TRIAL: NCT06990945
Title: Clinical Performance And Radiographic Assessment Of Mesoporous Bioactive Glass Adhesive Vs. Universal Adhesive In Class II Carious Lesions
Brief Title: The Study Aims to Compare the Effectiveness of Mesoporous Bioactive Glass-containing Adhesives vs Conventional Universal Adhesives on the Clinical Performance Composite Restorations Through Promoting Dentin Remineralization After Selective Caries Removal Over a Two-year Follow-up
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: providing support: Equipment and some consumables by Department of Oral Medicine, Periodontology and Oral Diagnosis, Faculty of Dentistry, Cairo University (Unknown)
Responsible Party: Principal Investigator, Ahmed Hesham samaha, PhD candidate Conservative Department Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU-2025-05; cu-fund-202505 (Other Grant/Funding Number: cairou)
Record Dates: First submitted 2025-05-08; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Dental Caries
Keywords: Class II Carious Lesions; Dentin Remineralization; Dental Adhesives; Bioactive Glass; Restorative Dentistry; Hypersensitivity
MeSH Terms: conditions — Dental Caries; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: the study is a 2-year, double-blind, randomized controlled trial with two parallel arms. Participants with Class II carious lesions will be randomly assigned to receive either a mesoporous bioactive glass adhesive (Hi-Bond Universal) or a conventional universal adhesive (OptiBond Universal). Clinical and radiographic assessments will be conducted at baseline, 6 months, 12 months, 18 months, and 24 months to evaluate the adhesive's performance in terms of fracture resistance, retention, marginal adaptation, dentin remineralization, and hypersensitivity.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study employs a double-blinded design to minimize potential biases in outcome assessment and data analysis. The following masking strategy will be implemented:
  Participant Blinding:
  Participants will be unaware of the type of adhesive used during the restorative procedure. Both adhesives (Hi-Bond Universal and OptiBond Universal) will be applied using identical clinical procedures to maintain blinding.
  Outcomes Assessor Blinding:
  The outcomes assessors (N.S. and R.A.), responsible for evaluating clinical performance (fracture resistance, marginal adaptation, hypersensitivity) and radiographic assessments, will be blinded to the group assignment. They will not have access to information regarding the type of adhesive used for each patient.
  Operator (A.H.) Not Blinded:
  The operator performing the restorative procedures cannot be blinded due to the nature of the intervention. The operator will be aware of the adhesive used but will not participate in the outcome assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Optibond Universal adhesive (Active Comparator): Participants in the control group will receive a conventional universal adhesive (OptiBond Universal) applied after selective caries removal. The adhesive will be applied according to the manufacturer's instructions, followed by placement of a nano-hybrid composite (Optishade Universal Kerr Dental).
  Interventions: Device: OptiBond Universal Adhesive
- Intervention - Hi-Bond Universal Adhesive (Experimental): Participants in this group will receive a bioactive glass-modified adhesive, Hi-Bond Universal (Mediclus, Korea). This adhesive releases calcium and phosphate ions to enhance dentin remineralization and reduce hypersensitivity, applied after selective caries removal and followed by composite restoration.
  Interventions: Device: Hi-Bond Universal Adhesive

INTERVENTIONS:
Device: Hi-Bond Universal Adhesive — A bioactive glass adhesive containing mesoporous bioactive glass designed to promote dentin remineralization, manufactured by Mediclus, Korea. It releases calcium and phosphate ions to enhance dentin sealing and reduce hypersensitivity
  The adhesive will be applied after selective caries removal following a standardized protocol:
  Selective enamel etching with 37% phosphoric acid for 15 seconds.
  Application of HI Bond Universal adhesive with agitation for 20 seconds.
  Light curing for 20 seconds using a LED curing device.
  Incremental application of a nano-hybrid composite (Optishade Universal Kerr Dental, USA).
  Occlusal adjustment, finishing, and polishing.
  Arms: Intervention - Hi-Bond Universal Adhesive
Device: OptiBond Universal Adhesive — conventional universal adhesive designed for bonding composite restorations to enamel and dentin.
  The adhesive will be applied after selective caries removal following a standardized protocol:
  Selective enamel etching with 37% phosphoric acid for 15 seconds.
  Application of OptiBond Universal adhesive with agitation for 20 seconds.
  Light curing for 20 seconds using a LED curing device.
  Incremental application of a nano-hybrid composite (Optishade Universal Kerr Dental, USA).
  Occlusal adjustment, finishing, and polishing.
  Arms: Optibond Universal adhesive

SUMMARY:
a two-year, double-blind, randomized controlled trial evaluates the effectiveness of a bioactive glass adhesive (Hi-Bond Universal) versus a conventional adhesive (OptiBond Universal) in Class II carious lesions. The study will assess clinical outcomes such as fracture resistance and marginal adaptation and radiographic evidence of dentin remineralization in 80 adult participants. Hypersensitivity and secondary caries development will also be monitored at multiple time points to determine comparative efficacy.

DETAILED DESCRIPTION:
This study is a two-year, double-blind, randomized controlled clinical trial designed to compare the clinical performance and radiographic outcomes of a mesoporous bioactive glass adhesive (Hi-Bond Universal) with a conventional universal adhesive (OptiBond Universal) in Class II carious lesions. The trial will enroll 80 participants aged 22 to 42 years, recruited from the Outpatient Clinic of the Conservative Dentistry Department at Cairo University.

Eligible participants presenting with ICDAS 5 and 6 carious lesions in posterior permanent teeth will be randomly assigned to one of two treatment groups. The intervention group will receive the Hi-Bond Universal adhesive, a bioactive glass-modified adhesive intended to promote dentin remineralization and reduce postoperative hypersensitivity through calcium and phosphate ion release. The control group will be treated with OptiBond Universal, a conventional adhesive providing mechanical bonding without bioactive properties.

Clinical outcomes will be evaluated using the FDI World Dental Federation criteria, focusing on functional properties such as fracture resistance, marginal adaptation, and retention. Radiographic assessments will quantify dentin remineralization using digital grayscale analysis. Hypersensitivity will be recorded using a patient-reported Likert scale at baseline, 6, 12, 18, and 24 months.

The primary outcome is the functional integrity of the restorative material, assessed at 24 months. Secondary outcomes include the presence of marginal caries, postoperative hypersensitivity, and radiographic evidence of dentin remineralization. Data will be analyzed using appropriate statistical methods to determine differences between the two adhesive systems.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 22 to 42 years.

Presence of Class II carious lesions in posterior permanent teeth (ICDAS 5 & 6).

Radiographic evidence of caries extending to 50% of dentin with a radiopaque layer between the lesion and pulp chamber.

Teeth with normal pulp vitality confirmed through cold pulp sensibility test.

Teeth with no periapical pathosis on radiographic examination.

Good oral hygiene as determined by the attending clinician.

Willingness to sign the informed consent and comply with the 2-year follow-up protocol.

Cooperative patients who can attend all follow-up visits.

Exclusion Criteria:

* Allergy to any of the restorative materials (OptiBond Universal or Hi-Bond Universal).

Patients currently undergoing orthodontic treatment with fixed appliances.

Pregnant women or those planning pregnancy during the study period.

Patients with systemic diseases that could interfere with dental treatment (e.g., uncontrolled diabetes, cardiovascular diseases).

Use of analgesics or medications that could mask postoperative sensitivity.

Teeth with previous restorations or treatment in the target area.

Teeth exhibiting spontaneous pain or lingering pain after sensitivity testing, indicating irreversible pulpitis.

Negative response in cold pulp sensibility test, indicating pulp necrosis.

Teeth with periapical radiolucencies or signs of infection.

Mobile teeth due to periodontal disease or trauma.

Teeth with extensive structural damage, such as cusp fractures or deep cracks.

Patients unable to comply with the follow-up schedule.

Ages: 22 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Performance - Functional Properties (Retention loss) | 24 months (Baseline, 6 months, 12 months, 18 months, 24 months)
  The clinical performance of the adhesive systems will be assessed based on the functional properties, specifically focusing on the retention of the composite Restoration Clinical assessment of the condition of adjacent mucosa to detect signs of irritation or inflammation caused by the adhesive materials.
  Assessment Method: FDI Criteria Scores (1-5)

SECONDARY OUTCOMES:
Clinical Performance - Functional Properties (fracture of the material) | 24 months (Baseline, 6 months, 12 months, 18 months, 24 months)
  Assessment of fracture resistance of the restorative materials (Hi-Bond Universal vs. OptiBond Universal) using the FDI Criteria. This includes the evaluation of material integrity, chipping, fractures, and overall structural durability of the restorations.Clinical assessment of the condition of adjacent mucosa to detect signs of irritation or inflammation caused by the adhesive materials.
  Assessment Method: FDI Criteria Scores (1-5)
Approximal Anatomical Form | 24 months (Baseline, 6 months, 12 months, 18 months, 24 months)
  Assessment of contact points and contours of the restoration, focusing on anatomical integrity and function.
  Assessment Method: FDI Criteria Scores (1-5)
Marginal Adaptation | 24 months (Baseline, 6 months, 12 months, 18 months, 24 months)
  Evaluation of the marginal adaptation of the adhesive systems using clinical criteria. This outcome assesses the adhesive's ability to seal restoration margins effectively.Clinical assessment of the condition of adjacent mucosa to detect signs of irritation or inflammation caused by the adhesive materials.
  Assessment Method: FDI Criteria Scores (1-5)
Clinical Performance - Biological Properties (Caries at Restoration Margins) | 24 months (Baseline, 6 months, 12 months, 18 months, 24 months)
  The presence of caries at restoration margins will be assessed using clinical examinations. The objective is to evaluate the adhesive's ability to prevent secondary caries development at the margins of the restorations.Clinical assessment of the condition of adjacent mucosa to detect signs of irritation or inflammation caused by the adhesive materials.
  Assessment Method: FDI Criteria Scores (1-5)
Postoperative Hypersensitivity | 24 months (Baseline, 6 months, 12 months, 18 months, 24 months)
  Assessment of patient-reported tooth hypersensitivity following adhesive application and composite restoration.Clinical assessment of the condition of adjacent mucosa to detect signs of irritation or inflammation caused by the adhesive materials.
  Assessment Method: FDI Criteria Scores (1-5)
Adjacent Mucosa Condition | 24 months (Baseline, 6 months, 12 months, 18 months, 24 months)
  Clinical assessment of the condition of adjacent mucosa to detect signs of irritation or inflammation caused by the adhesive materials.
  Assessment Method: FDI Criteria Scores (1-5)
Esthetic Properties - Staining (Surface and Margin) | 24 months (Baseline, 6 months, 12 months, 18 months, 24 months)
  Clinical evaluation of staining at the surface and margins of the restoration to assess esthetic integrity.
  Assessment Method: FDI Criteria Scores (1-5)
Remaining Dentin Bridge - Remineralization | 24 months (Baseline, 6 months, 12 months, 18 months, 24 months)
  Evaluation of remineralization at the remaining dentin bridge using digital radiography and grayscale analysis.
  Assessment Method: Digital Radiography (Grayscale values 0-255)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided